CLINICAL TRIAL: NCT03386266
Title: Biomarkers and Validation of Selected Outcome Measures (CMTNSmod)
Status: Completed | Type: Observational
Sponsor: University Medical Center Goettingen (Other)
Collaborators: University Hospital Muenster (Other); Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Michael W Sereda, MD, Professor of Neurology, Michael W Sereda, MD, Professor of Neurology, University Medical Center Goettingen
Other Study IDs: 05171
Record Dates: First submitted 2017-12-13; First posted 2017-12-29 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Charcot-Marie-Tooth Disease, Type IA
Keywords: Biomarkers; CMT1A; Charcot-Marie-Tooth disease
MeSH Terms: conditions — Charcot-Marie-Tooth Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA and RNA from blood and skin
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
CMT is a rare disease for which novel treatments are being developed. Evaluation of intervention efficacy is hampered by slow progression and lack of sensitive outcome measures. Primary goal of the project is to identify and validate RNA and protein derived biomarkers in blood of CMT patients for selected outcome measures over 2 years. The investigators expect to develop more responsive outcome measures and circulating biomarkers to improve assessment of intervention efficacy in forthcoming therapeutic trials.

DETAILED DESCRIPTION:
Novel treatments are being developed for CMT. Intervention efficacy evaluation is hampered by slow disease progression and lack of sensitive outcome measures. The investigators have previously shown that biomarkers from skin identified in a CMT1A rat model can be translated to CMT1A patients. Primary goal is to identify circulating biomarkers correlating with disease severity and progression. 210 young, adolescent and adult patients affected by genetically confirmed CMT1A, will be evaluated with different clinical outcome measures, assessing impairment, disability and quality of life: Patients will be re-evaluated at 12 (n=147) and 24 months (n=103) with the same measures to assess disease progression. A number of candidate markers correlating with disease severity have been identified in blood samples from the rat model of CMT1A. At 0-12-24 months a blood sample will be drawn from affected CMT1A patients. The investigators will purify total mRNA from blood samples, and validate the 10 strongest regulated markers identified in the rat model via qRTPCR in blood of CMT1A patients. Protein biomarkers will also be analysed. Marker expression at baseline and at follow up will be correlated with clinical severity and progression. In this translational project (rat/human) the investogators expect to develop more responsive outcome measures and circulating biomarkers to improve assessment of intervention efficacy in forthcoming therapeutic trials.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of CMT1A
* Genetic confirmation of PMP22 duplication (for adults patients)
* Children aged 3-11, adolescents aged 12-17 and adults aged 18-65 years
* Signed informed patient consent

Exclusion Criteria:

* Other causes of neurological and psychiatric disorders
* Severe internistic disease
* Patient known or suspected to be alcohol / drug abuser
* Pregnancy, breast feeding period
* Permanent Vitamin C intake
* Participation an interventional clinical study up to 4 weeks prior to inclusion

Ages: 3 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients suffering from CMT1A disease
Sampling Method: Non-Probability Sample
Enrollment: 156 (Actual)
Dates: Start 2017-08-11 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
mRNA Expression Levels in blood samples from CMT1A patients | 3 years
  Validation of key candidate genes (GSST2, FN3KRP, CTSA, SPRR1A) fro former studies
mRNA Expression Levels in Skin biopsies from CMT1A patients | 3 years
  Validation of key candidate genes (GSST2, FN3KRP, CTSA, SPRR1A) fro former studies

CONTACTS AND LOCATIONS:
Overall Officials: Michael W. Sereda, MD, Professor of Neurology, Principal Investigator — University Medical Center Goettingen
Locations (1):
- University Medical Center Goettingen, Goettigen, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mannil M, Solari A, Leha A, Pelayo-Negro AL, Berciano J, Schlotter-Weigel B, Walter MC, Rautenstrauss B, Schnizer TJ, Schenone A, Seeman P, Kadian C, Schreiber O, Angarita NG, Fabrizi GM, Gemignani F, Padua L, Santoro L, Quattrone A, Vita G, Calabrese D; CMT-TRIAAL/CMT-TRAUK Group; Young P, Laura M, Haberlova J, Mazanec R, Paulus W, Beissbarth T, Shy ME, Reilly MM, Pareyson D, Sereda MW. Selected items from the Charcot-Marie-Tooth (CMT) Neuropathy Score and secondary clinical outcome measures serve as sensitive clinical markers of disease severity in CMT1A patients. Neuromuscul Disord. 2014 Nov;24(11):1003-17. doi: 10.1016/j.nmd.2014.06.431. Epub 2014 Jun 19. PMID 25085517
- [Background] Fledrich R, Schlotter-Weigel B, Schnizer TJ, Wichert SP, Stassart RM, Meyer zu Horste G, Klink A, Weiss BG, Haag U, Walter MC, Rautenstrauss B, Paulus W, Rossner MJ, Sereda MW. A rat model of Charcot-Marie-Tooth disease 1A recapitulates disease variability and supplies biomarkers of axonal loss in patients. Brain. 2012 Jan;135(Pt 1):72-87. doi: 10.1093/brain/awr322. Epub 2011 Dec 20. PMID 22189569
- [Result] Fledrich R, Mannil M, Leha A, Ehbrecht C, Solari A, Pelayo-Negro AL, Berciano J, Schlotter-Weigel B, Schnizer TJ, Prukop T, Garcia-Angarita N, Czesnik D, Haberlova J, Mazanec R, Paulus W, Beissbarth T, Walter MC, Triaal C, Hogrel JY, Dubourg O, Schenone A, Baets J, De Jonghe P, Shy ME, Horvath R, Pareyson D, Seeman P, Young P, Sereda MW. Biomarkers predict outcome in Charcot-Marie-Tooth disease 1A. J Neurol Neurosurg Psychiatry. 2017 Nov;88(11):941-952. doi: 10.1136/jnnp-2017-315721. Epub 2017 Aug 31. PMID 28860329